CLINICAL TRIAL: NCT05152368
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cells Exosomes for the Treatment of Trigeminal Neuralgia
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Stem Cells Exosomes for Trigeminal Neuralgia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-1-MSC-019
Record Dates: First submitted 2021-11-29; First posted 2021-12-09 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Peripheral Neuropathy; Trigeminal Neuralgia
Keywords: Peripheral Neuropathy; Trigeminal Neuralgia; stem cell treatment
MeSH Terms: conditions — Peripheral Nervous System Diseases; Trigeminal Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (AlloEx) (Experimental): Intranasal installation of 4 CCs of AlloEx, which is approximately 800 billion exosomes.
  Interventions: Biological: AlloEx

INTERVENTIONS:
Biological: AlloEx — cultured allogeneic adult umbilical cord derived mesenchymal stem cell exosomes

SUMMARY:
This trial will study the safety and efficacy of instillation of cultured allogeneic adult umbilical cord derived mesenchymal stem cell exosomes for the treatment of Trigeminal Neuralgia.

DETAILED DESCRIPTION:
This patient funded trial aims to study the safety and efficacy of cultured allogeneic adult umbilical cord derived mesenchymal stem cell (UC-MSCs) exosomes for the treatment of Trigeminal Neuralgia. Patients will receive an intranasal instillation of UC-MSCs exosomes. The total dose will be approximately 800 billion exosomes split evenly between both nasal cavities via Tian Syringe through 4 CCs of AlloEx. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

For patients with more severe disease an autologous Effector cells (activated lymphocytes) treatment will be utilized created from the patient's own cells obtained by apheresis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Trigeminal Neuralgia or Peripheral Neuropathy
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (1):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda

IPD SHARING:
Plan to Share IPD: No